CLINICAL TRIAL: NCT02650986
Title: A Phase I/IIa Study of TGFß Blockade in TCR-Engineered T-Cell Cancer Immunotherapy in Patients With Advanced Malignancies
Brief Title: Gene-Modified T Cells With or Without Decitabine in Treating Patients With Advanced Malignancies Expressing NY-ESO-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I 258514; NCI-2015-02080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 258514 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); R01CA164333 (NIH)
Record Dates: First submitted 2015-12-21; First posted 2016-01-08 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Advanced Fallopian Tube Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Melanoma; Advanced Ovarian Carcinoma; Advanced Primary Peritoneal Carcinoma; Advanced Synovial Sarcoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Fallopian Tube Carcinoma; Metastatic Melanoma; Metastatic Ovarian Carcinoma; Metastatic Primary Peritoneal Carcinoma; Metastatic Synovial Sarcoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IIIA Fallopian Tube Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Primary Peritoneal Cancer AJCC v8; Stage IIIA1 Fallopian Tube Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Fallopian Tube Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Fallopian Tube Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Primary Peritoneal Cancer AJCC v8; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8; Unresectable Melanoma; Unresectable Ovarian Carcinoma; Unresectable Synovial Sarcoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Melanoma; Ovarian Neoplasms; Sarcoma, Synovial | interventions — Cyclophosphamide; Decitabine; Injections; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (cyclophosphamide, TCR/dnTGFbetaRII) (Experimental): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis; Biological: TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes
- Cohort II (decitabine, cyclophosphamide, TCR/dnTGFbetaRII) (Experimental): Patients undergo leukapheresis on day -6 and receive decitabine IV over 1 hour on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Interventions: Drug: Cyclophosphamide; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis; Biological: TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Cohort II (decitabine, cyclophosphamide, TCR/dnTGFbetaRII)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Biological: TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes — Given IV
  Other Names: TGFbDNRII-transduced Autologous TILs

SUMMARY:
This phase I/IIa trial studies the side effects and best dose of gene-modified T cells when given with or without decitabine, and to see how well they work in treating patients with malignancies expressing cancer-testis antigens 1 (NY-ESO-1) gene that have spread to other places in the body (advanced). A T cell is a type of immune cell that can recognize and kill abnormal cells of the body. Placing a modified gene for NY-ESO-1 into the patients' T cells in the laboratory and then giving them back to the patient may help the body build an immune response to kill tumor cells that express NY-ESO-1. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving gene-modified T cells with or without decitabine works better in treating patients with malignancies expressing NY-ESO-1.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of adoptive transfer of TGFbDNRII-transduced autologous tumor infiltrating lymphocytes (autologous NY-ESO-1 TCR/dnTGFbetaRII transgenic T cells).

SECONDARY OBJECTIVES:

I. NY-ESO-1 TCR/ dnTGFbetaRII transgenic T cell persistence by analyzing serial peripheral blood samples for the presence of T cells with the NY-ESO-1 TCR by tetramer analysis.

II. To study T cell differentiation that correlates with higher anti-tumor responses.

III. To test the hypothesis that NY-ESO-1 TCR/dnTGFbetaRII will constitute in cells more efficient in inducing tumor regression.

IV. Determine objective tumor responses by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) 1.1.

EXPLORATORY OBJECTIVE:

I. To evaluate the role of microbiota on the therapeutic efficacy of the proposed therapy.

OUTLINE: This is a phase I, dose-escalation study of NY-ESO-1 TCR/TGFbDNRII-transduced TILs followed by a phase IIa study. Participants are assigned 1 to 2 cohorts.

COHORT I: Patients undergo leukapheresis on day -6, and receive cyclophosphamide intravenously (IV) over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.

COHORT II: Patients undergo leukapheresis on day -6 and receive decitabine IV over 1 hour on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.

After completion of study treatment, patients are followed up at weeks 1-4, 6, 8, and 12, at 6 and 9 months, every 6 months for 5 years, and then yearly for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors as described below:

  * Inoperable or metastatic (advanced) melanoma:

    * Has received, is intolerant, or refused a CTLA-4 inhibitor (ipilimumab) or a PD-1 inhibitor (nivolumab or pembrolizumab) as monotherapy and/or a combination of ipilimumab and nivolumab
    * Has received or is intolerant of a BRAF inhibitor or the combination of BRAF and MEK inhibitors for BRAFv600 mutant melanoma and a PD-1 inhibitor as monotherapy or in combination
  * Inoperable or metastatic (advanced) ovarian, primary peritoneal or fallopian tube carcinoma:

    * Has received platinum containing chemotherapy and has platinum refractory or resistant disease that has progressed on second line therapy
    * If platinum sensitive disease, should have received >= 2 lines of chemotherapy
    * May have received PARP inhibitors, bevacizumab or other targeted VEGF inhibitor therapy
  * Inoperable or metastatic (advanced) synovial sarcoma:

    * Should have received and progressed on >= two lines of systemic therapy
  * Subjects with other histologies:

    * Must have previously received two lines of systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been deemed either non-responders (progressive disease) or have recurred
* For cohorts 1, 2 and 3 only: Patient's tumor must be positive by histological or molecular assay for NY-ESO-1, according to the screening algorithm; historical results may be used

  * For cohort 4, NY-ESO-1 results will be noted but NY-ESO-1 positivity is not required for eligibility
* Human leukocyte antigen (HLA)-A*0201 (HLA-A2.1) positivity by molecular subtyping (blood test or buccal swab, historical documentation acceptable)
* Age >= 18 years old, (Cohort 4: Age >= 12 years old)
* Life expectancy greater than 3 months assessed by a study physician
* Have been informed of other treatment options
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to irRECIST criteria
  * For patients with skin metastases, lesions selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s)
* No restriction based on prior treatments but at least 4 weeks from prior immunotherapy, or prior investigational agents. Note: Patients who have suffered >grade 2 irAEs during previous checkpoint inhibitor therapy should be excluded.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Must have adequate venous access for apheresis
* Women of childbearing potential and men must agree to use effective methods of birth control for the duration of the study and 6 months after; methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception; it is recommended that a combination of two methods be used
* Leukocytes: >= 3,000/mcl
* Absolute neutrophil count: >= 1,000/mcl
* Platelets: >= 100,000/mcl
* Total bilirubin: =< 1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): =< 2.5 x institutional upper limit of normal
* Creatinine: =< 2 X ULN; if creatinine > 2 X ULN, creatinine clearance must be > 60 ml/min
* Must be willing and able to accept the leukapheresis procedure
* At screening, must have tissue available for NY-ESO-1 testing (if not previously performed) or be willing and able to undergo a fresh tissue biopsy
* Patient must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participant must agree to and arrange for a caregiver (age >= 18 years old) available 24 hours a day/ 7 days a week and arrange for lodging within 45 minutes drive to Roswell Park and transportation for a period of time after discharge from the hospital; the exact amount of time will depend on the individual status as determined by the treating physician
* ELIGIBILITY CRITERIA FOR A SECOND TRANSGENIC T CELL INFUSION

Subjects in whom disease control was observed after the T cell infusion may be eligible for a second transgenic T cell infusion if the subject meets the following criteria:

* Patient attained confirmed disease control (either complete remission [CR], partial remission [PR] or stable disease [SD]) after the first transgenic T cell infusion
* Patient still meets the eligibility criteria above
* A second T cell infusion is discussed and the patient agrees to receive it
* Either cryopreserved extra cells from the first T cell product is available or cryopreserved autologous peripheral blood mononuclear cell (PBMC) is available for the manufacture of a second transgenic T cell product

Exclusion Criteria:

* Previously known hypersensitivity to any of the agents used in this study
* Currently receiving any other investigational agents. Note: Patients who have suffered >grade 2 irAEs during previous checkpoint inhibitor therapy should be excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; electrocardiogram (EKG) will be done at screening; cardiac stress test will be done as clinically indicated, the specific test to be chosen at the discretion of the treating physician.
* History of severe autoimmune disease requiring steroids or other immunosuppressive treatments
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, which in the investigator's opinion would place the patient at an increased risk for adverse effect or current acute colitis of any origin; treated cases with no active disease are eligible
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 4 weeks prior to enrollment (inhaled or topical steroids at standard doses or isolated use of steroids as premedication for medical procedures to minimize allergic reaction [e.g. computed tomography (CT) scan dye] are allowed)
* Known active infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C or cytomegalovirus (CMV)
* Known cases of clinically active brain metastases (brain magnetic resonance imaging [MRI] as clinically indicated); prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of compliance with the requirements of this protocol even with caregiver support
* Pregnancy or breast-feeding; female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and 6 months after; all female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 48 hours from starting the conditioning chemotherapy
* Lack of availability of a patient for immunological and clinical follow-up assessment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2032-07-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philip McCarthy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV at 1 x 10^7
- Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV at 1 x 10^8
- Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV at 1 x 10^9
- Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3): Patients undergo leukapheresis on day -6 and receive decitabine IV over 1 hour on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV
  Decitabine: Given IV at 20 mg/m^2 x 3 days
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV at 1 x 10^9
Period: Overall Study
Arm/Group | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3)
Started | 3 | 3 | 3 | 6
Completed | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3): Patients undergo leukapheresis on day -6 and receive decitabine IV over 1 hour on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV at 1 x 10^9
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 2 | 3 | 3 | 5 | 13
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Year] | 62.2 (8.3) | 61.4 (2.0) | 60.1 (2.7) | 43.8 (18.4) | 54.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 8
  Male | 1 | 0 | 2 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Will be assessed using Common Toxicity Criteria. Patients will be monitored by medical histories, physical examinations, ophthalmologic exams, and blood studies to detect potential toxicities from the treatment.
  the number of patients experiencing a DLT are reported.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV at 1 x 10^7
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV
- Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV at 1 x 10^8
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV
- Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3): Patients undergo leukapheresis on day -6 and receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV at 1 x 10^9
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
  TGFbDNRII-transduced Autologous Tumor Infiltrating Lymphocytes: Given IV
- Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3): Patients undergo leukapheresis on day -6 and receive decitabine IV over 1 hour on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then receive TGFbDNRII-transduced autologous tumor infiltrating lymphocytes IV over 15 minutes on day 0. Eligible patients who showed initial response/disease control, may receive a second TGFbDNRII-transduced autologous tumor infiltrating lymphocytes infusion at any time after progression is confirmed.
  Cyclophosphamide: Given IV at 1 x 10^9
  Decitabine: Given IV at 20 mg/m^2 x 3 days
  Laboratory Biomarker Analysis: Correlative studies
  Leukapheresis: Undergo leukapheresis
Arm/Group | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3)
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Feasibility Concerns in Manufacturing of NY-ESO-1/ dnTGFbetaRII Engineered Cells
Description: Unfeasibility will be defined as 3 or more preparations not meeting the lot release criteria in each cohort. Sufficient numbers of circulating, lot released confirmed T cells will be measured prior to administration.
  The count of patients not meeting the preparation criteria are reported.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3)
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 1 | 0 | 0

3. Secondary Outcome: Expression of the NY-ESO-1 T Cell Receptor (TCR) Transgenic Protein in Peripheral Blood Mononuclear Cells (PBMC)
Description: TCR and vector presence will be quantitated in PBMC samples, obtained before adoptive transfer and at weeks 1, 2, 4, 8, and 12 after transgenic cell adoptive transfer. Thereafter, sampling will be every 3 months during the first year, and then every 6 to 12 months per schedule of procedures and observations.
Time Frame: Up to 15 years
Reporting Status: Not Posted

4. Secondary Outcome: Replication Competent Retrovirus (RCR)
Description: Will be assessed in blood by polymerase chain reaction (PCR).
Time Frame: Up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Tumor Response (Complete and Partial Response)
Description: Will be determined by immune-related Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Response assessment will be performed by comparing standard computed tomography imaging scans and photographs of target lesions from baseline.
Time Frame: Up to 90 days after TCR transgenic PBMC adoptive transfer
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were captured during treatment and up to 30 days post treatment. Based on the observed data, the AE time frame was from 1.1 to 22.3 months.
Arm/Group | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 2/3 | 4/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) (N=3) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) (N=3) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) (N=3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Chills (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 3 (9) | 0 (0) | 1 (4)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 1) (N=3) | Cohort 2 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 2) (N=3) | Cohort 3 (Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) (N=3) | Cohort 4 (Decitabine, Cyclophosphamide, TCR/dnTGFbetaRII - Dose Level 3) (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (18) | 1 (3) | 2 (18) | 4/5 (40)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (12) | 1/5 (8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (8)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Abdominal hernia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 1 (15) | 0 (0) | 0/5 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (6) | 1/5 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 2 (9) | 1/5 (4)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 1 (3) | 0 (0) | 0/5 (0)
Dysphagia (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0/5 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Nausea (Gastrointestinal disorders) | 1 (8) | 2 (6) | 2 (9) | 3/5 (24)
Oesophagitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Stomatitis (Gastrointestinal disorders) | 1 (6) | 0 (0) | 1 (3) | 0/5 (0)
Vomiting (Gastrointestinal disorders) | 2 (6) | 3 (9) | 2 (12) | 1/5 (4)
Asthenia (General disorders) | 1 (3) | 0 (0) | 1 (3) | 0/5 (0)
Catheter site pain (General disorders) | 1 (3) | 1 (3) | 0 (0) | 0/5 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1/5 (4)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Face oedema (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0/5 (0)
Fatigue (General disorders) | 3 (12) | 2 (18) | 2 (6) | 1/5 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Localised oedema (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Medical device pain (General disorders) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Oedema (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Oedema peripheral (General disorders) | 3 (14) | 2 (9) | 1 (3) | 0/5 (0)
Pain (General disorders) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (6) | 2/5 (8)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Cytokine release syndrome (Immune system disorders) | 1 (3) | 0 (0) | 0 (0) | 3/5 (12)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0/5 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Herpes zoster (Infections and infestations) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Rhinitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (3) | 0/5 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 0 (0) | 1 (6) | 0/5 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Blood creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Brain natriuretic peptide increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Cardiac murmur (Investigations) | 1 (3) | 1 (3) | 0 (0) | 0/5 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2/5 (12)
Neutrophil count decreased (Investigations) | 2 (9) | 1 (9) | 0 (0) | 2/5 (12)
Neutrophil count increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Platelet count decreased (Investigations) | 2 (18) | 0 (0) | 0 (0) | 2/5 (24)
Platelet count increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
White blood cell count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
White blood cell count decreased (Investigations) | 3 (26) | 2 (6) | 0 (0) | 3/5 (56)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (3) | 0/5 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 0 (0) | 0/5 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1/5 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 3/5 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1/5 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (8)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (12) | 0 (0) | 2 (6) | 0/5 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (3) | 1 (3) | 1/5 (4)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Dizziness (Nervous system disorders) | 2 (8) | 1 (3) | 0 (0) | 1/5 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Headache (Nervous system disorders) | 2 (11) | 1 (6) | 0 (0) | 2/5 (8)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0/5 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Mental status changes (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 1/5 (4)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (6) | 0/5 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (6) | 0 (0) | 0/5 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (11) | 1 (3) | 0 (0) | 0/5 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (6) | 0/5 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 2/5 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1/5 (8)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0/5 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0/5 (0)
Hypertension (Vascular disorders) | 1 (15) | 0 (0) | 0 (0) | 0/5 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (6) | 1/5 (4)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0/5 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02650986/Prot_SAP_000.pdf